CLINICAL TRIAL: NCT05569746
Title: A Phase II Study to Assess Safety, Efficacy, and Pharmacokinetics of INM004 (Anti-Shiga Toxin) in Pediatric Patients With Hemolytic Uremic Syndrome Associated With Shiga Toxin-producing Escherichia Coli Infection
Brief Title: A Study to Assess Safety, Efficacy, and Pharmacokinetics of INM004 in Pediatric Patients With STEC-HUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inmunova S.A. (Other)
Collaborators: KLIXAR (Unknown); Linical Co., Ltd. (Industry); PHV LATAM (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-INM004-03
Record Dates: First submitted 2022-08-22; First posted 2022-10-06 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2022-10

CONDITIONS: Diarrhea-Associated Hemolytic Uremic Syndrome; Pediatric Kidney Disease; Hemolytic-Uremic Syndrome
Keywords: STEC-HUS
MeSH Terms: conditions — Hemolytic-Uremic Syndrome

STUDY DESIGN:
Intervention Model Description: A Phase II, multicenter, controlled study, with a prospective open "treatment group" (with INM004 added to Standard of Care) and a retrospective "control group" (only treated with Standard of Care).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INM004 (Experimental): 2 doses of 4 mg/kg separated by 24 h
  Interventions: Drug: INM004; Other: SoC

INTERVENTIONS:
Drug: INM004 — Two 4 mg/kg doses of INM004, 24 h (±2 h) apart, will be assessed. Each dose will be administered as an intravenous infusion during 50 min.
  Other Names: Equine immunoglobulin fragment F(ab')2 anti-Shiga toxin
Other: SoC — Standard of care

SUMMARY:
Hemolytic Uremic Syndrome (HUS) is a foodborne disease which mainly affects children. It is caused by Escherichia coli bacteria, which release a toxin called Shiga toxin within the body. This infectious form of HUS, defined as STEC-HUS, can cause sporadic cases or outbreaks, as observed in different countries. Argentina has the highest incidence of STEC-HUS worldwide. The disease is endemic, representing approximately 95% of all HUS cases nationwide.

STEC-HUS generally begins with diarrhea (with or without blood), and can also cause fever, abdominal pain, and cramps. Then the child may have pallor, altered consciousness, decreased urine output, seizures, and other symptoms. Although death is uncommon (it occurs in 2-4% of cases), it is a very serious disease that mainly affects the kidneys, and also other organs such as the brain. About half of children need to undergo a risky procedure such as dialysis (due to malfunctioning kidneys); and most of them also receive blood transfusions.

Around 30% of the patients are left with lifelong consequences that can range from permanent kidney damage to the need for a transplant.

So far there is no drug, antibiotic or vaccine to prevent or treat HUS. Current treatment protocols include hospitalization for all patients with HUS, and supportive therapy such as hydration and salt intake. Support therapy is not a specific treatment, but rather helps the body better defend itself against the disease.

The purpose of this study is to establish whether it is safe and effective to treat patients who are diagnosed with STEC-HUS, with INM004 (study drug). INM004 is an investigational product "Fraction F(ab')2 of Equine Shiga Antitoxin Immunoglobulin". It is a concentrated and sterile serum obtained from healthy horses immunized against Shiga toxin that contains antibodies capable of neutralizing it.

The initial hypothesis is that INM004 would neutralize the entry of Shiga toxin into the body's cells thus preventing the consequent toxic damage. With the proposed treatment, INM004 would eliminate the Shiga toxin, preventing the progression of HUS symptoms and its serious complications (such as the need for and duration of dialysis, duration of hospital stays, as well as neurological, cardiovascular, intestinal complications, among others) which are associated with high morbidity and mortality. This treatment could then have an impact in health costs of STEC-HUS as well as the social costs.

DETAILED DESCRIPTION:
Hemolytic uremic syndrome (HUS) is a form of thrombotic microangiopathy characterized by microangiopathic hemolytic anemia, thrombocytopenia, and acute renal failure. HUS of infectious origin, associated with infection by Shiga toxin (Stx)-producing Escherichia coli.

This disease can cause sporadic cases or outbreaks. Argentina is the country with the highest incidence of STEC-HUS worldwide. The disease is endemic, representing approximately 95% of all HUS cases.

There is no specific treatment capable of preventing or controlling renal and extrarenal damage caused by Stx. The treatment is mainly symptomatic. Therapy for patients with acute kidney injury is supportive and includes hydric and electrolyte management; thus, most cases require red blood cell transfusions and approximately half of cases require dialysis.

INM004 is a neutralizing serum consisting of the F(ab')2 fragment of equine immunoglobulins with specificity against the B subunits of Stx1 and Stx2. The F(ab')2 fragments are obtained through the processing of serum from horses immunized with Stx1B and Stx2B immunogens, obtained through genetic engineering techniques. A polyclonal therapy based on INM004 offers the advantage that the different subtypes of Stx could be recognized by multiple antibodies simultaneously, even when the toxin circulates bound to neutrophils or microvesicles derived from them.

The objective of this study is to evaluate the efficacy, safety, and pharmacokinetics of INM004 administered in patients between 1 and 12 years of age who are in the early stage of the disease.

The initial hypothesis is that INM004 would reduce the complications associated with STEC-HUS by neutralizing the harmful effect of Stx on the body. Intravenous administration of INM004 is expected to interrupt the Stx-mediated cascade, reducing the occurrence of renal and extrarenal complications (such as the need for and duration of dialysis, number of transfusions, CNS complications, and length of hospitalization).

Two doses of 4 mg/kg of INM004 will be administered as an intravenous infusion over a period of 50 min, with an interval of 24 h (± 2 h) from each other. The selection of the exposure level is based on preclinical in vitro data regarding the affinity of INM004, its neutralizing capacity for both Stx toxins, and clinical data obtained from the previous Phase I study in adult volunteers and the Phase 2/3 study in children with STEC bloody diarrhea.

Study design: A Phase II, multicenter, controlled study, with a prospective open "treatment group" (with INM004 and Standard of Care -SoC-), and a retrospective "control group" (only treated with SoC). Considering that STEC-HUS is an orphan disease currently without treatment, the design with retrospective control has been chosen.

The treatment group will enroll 100 patients hospitalized in 16 healthcare centers in Argentina, between September 2022 and May 2023, time of highest incidence of STEC-HUS. The data of the control group will be obtained retrospectively from 200 cases of STEC-HUS treated in the same centers, in the same seasonal period in the years 2018, 2019 and until March 2020 (COVID-19 pre-pandemic), with the same screening criteria as the subjects in the treatment group.

Primary Objectives: To assess: 1) the efficacy of INM004, plus SoC, in the treatment of STEC-HUS, in terms of improvement of renal involvement; 2) the safety of the administration of INM004; 3) the pharmacokinetics (PK) of INM004.

Secondary Objectives: To assess the efficacy of INM004: 1) in the mortality reduction; 2) in the improvement of the STEC-HUS associated thrombotic microangiopathy, plus SoC; 3) in the treatment of STEC-HUS, in the prevention and reduction of renal involvement in the short term, plus SoC; 4) in the treatment of STEC-HUS, in the prevention and reduction of extrarenal involvement in the short term, plus SoC; 5) the in the prevention and reduction of the complications not associated to thrombotic microangiopathy, plus SoC; 6) in terms of the length of hospital stay; and 7) the evolution of laboratory parameters of interest after the administration of INM004.

Exploratory Objectives: To assess: 1) the immunogenicity of INM004; 2) the presence of circulating Stx before the administration of INM004; 3) the immune response to STEC infection over 4 weeks follow-up; 4) the correlation between serotype/ genotype of isolated STEC strains and disease severity.

Study Procedures:

For the control group: Data will be collected from the medical records of the subjects who have been eligible from the "Potential Subjects Selection List" of the year's corresponding to this population. The data to be collected for this group will be the same as for the treatment group, except for that related to the specific procedure of the intervention: basal ECG and post dose control; 1st dose and 2nd dose, and associated controls (vital signs and AESI evaluation); blood samples for biological and/or pharmacokinetic studies; adverse events.

The inclusion of subjects in the treatment group will be conducted in two stages: Stage 1 (Safety): A safety analysis will be performed by the Data Safety Monitoring Board (DSMB) after the first 12 subjects have been enrolled and 24 h after the administration of the second dose of INM004 have occurred. Stage 2 (Safety and Efficacy): Enrollment will continue until May 2023, and it is estimated that 88 more subjects will enroll in this stage.

Once the participant was included the following data will be collected:

Demographic data, medical history data, data of the current illness (related to the prodromal period of STEC-HUS and to the clinical features compatible with STEC-HUS at the time of diagnosis); Complications associated with STEC-HUS at the time of diagnosis and before: renal, neurological, cardiovascular, gastrointestinal, endocrinological, hematologic, lung involvement, infectious compromise. The follow up will continue to the day 28 after diagnosis.

For statistical analyses, the following populations will be considered:

* Full Analysis Set (FAS): For the treatment group, defined as all subjects who received at least 1 dose of INM004 with available follow-up evaluation on at least one efficacy parameter. This population will be used for all main efficacy analyses. All subjects included in the control group will be part of the FAS for the comparative analyses.
* Population by Correct Protocol (PCP): includes all the subjects in the FAS who did not present major deviations from the protocol that could affect the measures of efficacy. This population will be analyzed as a sensitivity evaluation for the main analyzes of the study.
* Safety Population (SP): For the treatment group, it is defined as all subjects who have received at least one dose of INM004.

Statistical methods:

Statistical analyzes will be mainly descriptive. For continuous variables, mean, median, standard deviation, quartiles, maximum and minimum will be presented. Categorical variables will be described by absolute frequencies and percentages.

Baseline parameters, demographics, clinical history and previous treatments will be described in a cross-sectional manner prior to the start of treatment. The continuous evaluations carried out throughout the study will be described longitudinally by the change from baseline. For categorical variables, shift tables can be generated.

In the treatment group, the last measure performed prior to the administration of the first dose of INM004 will be considered as the baseline measure of efficacy and safety. If a generalized delay in the administration of the INM004 treatment is observed, the closest measurement available to the diagnosis of symptoms compatible with STEC-HUS may be considered as the baseline measurement. For the control group, the baseline assessments will be those at the time of diagnosis of symptoms compatible with STEC-HUS.

Multivariate analyzes will be assessed to identify risk factors related to the evolution and severity of the disease.

Safety will be assessed throughout the study describing subjects with at least one AE, serious adverse events (SAE) and AESI, and subjects with at least one major safety deviation for each of the parameters: ECG, vital signs, clinical laboratory evaluations, including liver function tests.

Efficacy and sensitivity analyzes will be performed to detect possible subjects who could benefit more from treatment in subgroups defined according to levels of severity at admission Comparative multivariate analyzes of the main efficacy variables against the control group will be performed. These comparisons will be duly adjusted using propensity scoring techniques in order to minimize any confusion bias between both groups. Among the potential confounders to consider as adjustment variables in the model will be age, sex and severity levels at admission. Due to the exploratory nature of the comparisons, no adjustments will be made for multiple comparisons.

Due to the exploratory nature of this study, a sample of approximately 100 evaluable subjects in the treatment group would be sufficient to detect any existing trends regarding the efficacy and safety of INM004. In the control group, 200 subjects are expected to be evaluated.

With 100 evaluable subjects we will obtain a precision (distance from the mean to the end of the bilateral confidence interval at 95%) of ±1.2 for the days on dialysis (SD 6.1 days) and ±2.4 for the days of admission (SD 12 days).

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥1 and <12 years.
2. With hospitalization criterion in the participating facility.
3. Clinical event with a diagnosis compatible with STEC-HUS defined as:

   1. Presence of signs of kidney injury defined as:

      * Serum creatinine value above the UNL for age and sex, and/or
      * Hematuria (≥5 red blood cells per field or ≥27 red blood cells/μL in urine sediment),
   2. And at least 1 of the following 2 criteria:

      * Presence of hemolysis documented by: LDH levels above the UNL for age, and/or presence of schistocytes in peripheral blood smears.
      * Platelet consumption according to any of the following laboratory criteria: Platelet count <150 × 103/μl, in peripheral blood, and/or ≥50% decrease in peripheral blood platelet count compared to the baseline sample or within the previous 24 h.
4. Onset of diarrhea no more than 13 days at the time of diagnosis of a condition compatible with STEC-HUS at the participating facility.
5. For the treatment group, informed consent form signed and dated by the parent(s) or legal guardian with the assent of the subject as appropriate based on age and regulatory guidelines.
6. For the treatment group, female girls/adolescents who are already fertile must have a negative pregnancy test. Note: They will be considered fertile when they have already had menarche.

Exclusion Criteria:

1. With dialysis for more than 48 h at the time of diagnosis of a condition compatible with STEC-HUS in the participating facility.
2. History of chronic/recurrent hemolytic anemia, thrombocytopenia, or chronic renal failure.
3. Personal and/or family history of atypical HUS.
4. Suspected HUS secondary to other infectious processes not from gastrointestinal origin.
5. Evidence of clinically significant chronic active disease that is not medically controlled whose symptoms/signs may interfere with the treatment/diagnosis of this study, in the opinion of the investigator.
6. For the interventional group, history of: a) anaphylaxis of any type; b) previous administration of equine serum (for example, anti-venom serum, anti-spider toxin serum, anti-SARS-CoV-2 serum, etc.) or an allergic reaction from contact or exposure to horses.
7. Pregnant or lactating women.
8. For the interventional group, the impossibility of hospitalization in the participating institution.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Days of dialysis | 28 days
  Days of dialysis recorded as a continuous variable from 0 to 28 days
Adverse events (AEs) | 28 days
  Incidence of AEs classified according to affected organ systems and according to severity Incidence of AEs of special interest: incidence of injection site reactions and hypersensitivity reactions (ie, allergic reaction, anaphylaxis, and serum sickness).
Pharmacokinetics (PK) Evaluation of INM004 | 0, 1, 24, 26, 48 and 120 hours post-dose
  Serum concentration of INM004 at different time intervals in subjects participating in this substudy

SECONDARY OUTCOMES:
Mortality | 28 days
  Number of participants who survive after 4 weeks of follow-up
Change in thrombotic microangiopathy involvement (Creatinine %) | 28 days
  Percentage of subjects with normalization and/or stabilization for Creatinine
Change in thrombotic microangiopathy involvement (Creatinine) | 28 days
  Days until normalization and/or stabilization for Creatinine
Change in thrombotic microangiopathy involvement (Hematuria %) | 28 days
  Percentage of subjects with normalization and/or stabilization for Hematuria
Change in thrombotic microangiopathy involvement (Hematuria) | 28 days
  Days until normalization and/or stabilization for Hematuria
Change in thrombotic microangiopathy involvement (Proteinuria %) | 28 days
  Percentage of subjects with normalization and/or stabilization for Proteinuria
Change in thrombotic microangiopathy involvement (Proteinuria) | 28 days
  Days until normalization and/or stabilization for Proteinuria
Change in thrombotic microangiopathy involvement (GFR) | 28 days
  Days until normalization and/or stabilization for glomerular filtration rate
Change in thrombotic microangiopathy involvement (GFR %) | 28 days
  Percentage of subjects with normalization and/or stabilization for glomerular filtration rate
Change in thrombotic microangiopathy involvement (LDH %) | 28 days
  Percentage of subjects with normalization and/or stabilization for LDH
Change in thrombotic microangiopathy involvement (LDH) | 28 days
  Days until normalization and/or stabilization for LDH
Change in thrombotic microangiopathy involvement (Platelet) | 28 days
  Days until normalization and/or stabilization for platelet
Change in thrombotic microangiopathy involvement (Platelet %) | 28 days
  Percentage of subjects with normalization and/or stabilization for platelet
Change in thrombotic microangiopathy involvement (Hemoglobin %) | 28 days
  Percentage of subjects with normalization and/or stabilization for Hemoglobin
Change in thrombotic microangiopathy involvement (Hemoglobin) | 28 days
  Days until normalization and/or stabilization for Hemoglobin
Change in renal involvement (dialysis) | 28 days
  Assessed as a dichotomous variable (yes/no)
Change in renal involvement (dialysis subgroups) | 28 days
  Assessed as an ordinal variable (subjects without dialysis, with dialysis between 1-10 days, and subjects with dialysis >10 days).
Change in renal involvement (anuria) | 28 days
  Days of anuria (diuresis < 0.5 ml/kg/d)
Change in renal involvement (hypertension) | 28 days
  Number of participants with hypertension
Change in extrarenal involvement (hematological Interventions) | 28 days
  Number of participants with Requirement for red blood cell transfusions, Requirement for platelet transfusions
Change in extrarenal involvement (hematological Clinical) | 28 days
  Number of participants with Petechiae and/or bruising.
Change in extrarenal involvement (neurological) | 28 days
  Number of participants with Impaired consciousness, Seizure, Focal deficit
Change in extrarenal involvement (cardiovascular) | 28 days
  Number of participants with Cardiovascular instability, Acute myocardial infarction, Myocarditis, Arrhythmia
Change in extrarenal involvement (gastrointestinal) | 28 days
  Number of participants with Hemorrhagic colitis, Ischemic colitis, Bowel perforation, Intussusception, Pancreatitis, Hepatitis, Ilium
Change in extrarenal involvement (endocrine) | 28 days
  Number of participants with Hyperglycemia with insulin requirement
Change in secondary complications (pulmonary) | 28 days
  Number of participants with Pulmonary edema, Respiratory distress syndrome
Change in secondary complications (infectious involvement) | 28 days
  Number of participants with Peritonitis, Urinary tract infection, Bacteremia, Abscesses
Change in the length of hospital stay | 28 days
  Days of hospital stay (between hospital admission and discharge)
Change in laboratory parameters associated with worse prognosis | 28 days
  Changes in values of laboratory parameters of interest

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Goldbaum, PhD, Study Director — Inmunova S.A.
Locations (16):
- Argentina (16):
  - Hospital Interzonal Dr. José Penna, Bahía Blanca, Buenos Aires
  - Hospital De Niños Sor María Ludovica, La Plata, Buenos Aires
  - Hospital Interzonal Especializado Materno Infantil Don Victorio Tetamanti, Mar del Plata, Buenos Aires
  - Hospital El Cruce - Néstor Kirchner, San Juan Bautista, Buenos Aires
  - Hospital Dr. Lucio Molas, Santa Rosa, La Pampa Province
  - Sanatorio de Niños, Rosario, Santa Fe Province
  - Hospital General de Niños Pedro de Elizalde, Buenos Aires
  - Clínica Zabala Swiss Medical, Buenos Aires
  - Hospital de Pediatría Garrahan, Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma de Buenos Aire
  - Hospital de Niños Dr. Ricardo Gutierrez, Ciudad Autonoma de Buenos Aire
  - Sanatorio Güemes, Ciudad Autonoma de Buenos Aire
  - Hospital de Niños de la Santísima Trinidad, Córdoba
  - Sanatorio Allende, Córdoba
  - Hospital Pediátrico Dr. Humberto Notti, Mendoza
  - Hospital Provincial Neuquén Dr. Eduardo Castro Rendón, Neuquén

IPD SHARING:
Plan to Share IPD: No